CLINICAL TRIAL: NCT01270685
Title: 2009 H1N1 Pandemic and Seasonal Influenza in SCI/D: Infection Control Strategies
Status: Withdrawn | Type: Observational
Why Stopped: Not a Clinical Trial requirement per VA HSR&D
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: LaVela, Sherri - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: RRP 10-046
Record Dates: First submitted 2010-06-03; First posted 2011-01-05 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Veterans with spinal cord injuries and disorders
- 2: Comparison group: general Veteran population (without spinal cord injuries or disorders)
- 3: Health care providers with face-to-face contact with Veterans with SCI/D
- 4: Infection control Chiefs/Officers

SUMMARY:
The purpose of this study is to evaluate specific approaches used to prevent/reduce influenza transmission in the SCI/D System of Care in response to the 2009 H1N1 pandemic, including assessing infection control strategies used by SCI staff and guidance provided by local infection control units. Due to the rapid spread of and uncertainties about the H1N1 virus, we will evaluate patient's beliefs, behaviors, and information seeking strategies (e.g., social media). These findings will lend to the understanding of ways to handle emergent issues, such as the H1N1 pandemic, in special populations.

DETAILED DESCRIPTION:
In the United States, H1N1 influenza has been widespread, resulting in many infections, hospitalizations, and deaths. Due to impaired respiratory function following injury, persons with spinal cord injuries and disorders (SCI/D) are at extremely high risk from respiratory complications that occur as a result of contracting influenza.

The overall goal is to understand approaches used to prevent/reduce influenza transmission in the SCI/D System of Care in response to the 2009 H1N1 pandemic, in addition to seasonal influenza. Due to the rapid spread of and uncertainties about the H1N1 virus, one objective is to evaluate patient's beliefs, behaviors, and information seeking strategies (e.g., social media). The other objective is to assess infection control strategies used by SCI staff (and perceptions of) and guidance provided by local infection control units.

Multiple data collection efforts will be used to evaluate strategies used and their impact to address influenza (H1N1 and seasonal) in the VHA SCI/D population. At the facility level, the guidance provided by local infection control units in general and specific to SCI/D will be assessed via a semi-structured interview with infection control Chiefs/liaisons. An anonymous survey will be conducted to assess SCI health care providers' beliefs about and use of infection control strategies (vaccination and non-vaccine methods such as personal protective equipment, hand hygiene practices, appropriate work attendance practices) in addition to their perceptions of strength of evidence for H1N1 prevention measures, resource availability, and outreach by local infection control to facilitate infection prevention strategies. In addition, Veterans with SCI/D will be surveyed about their beliefs and information seeking strategies (e.g., social media) about seasonal and H1N1 influenza during the most recent influenza season, in addition to occurrence of influenza/ILI, receipt of influenza vaccination (H1N1 and/or seasonal) during the current influenza vaccination period, and perceived adverse effects from vaccination. Finally, the use of antiviral medications to treat influenza in Veterans with SCI/D, a two-group retrospective pre-posttest review of all visits and admissions associated with influenza (or related) diagnosis and/or antiviral prescription will be conducted. Charts for Veterans with SCI/D and Veterans who do not have SCI/D will be reviewed and compared for differences in practices in the SCI/D population versus the general veteran population.

This study will provide critical information that can be used to improve compliance with and understanding of influenza vaccination and infection control strategies at the patient, provider, and facility levels. These findings will lend to the understanding of ways to handle emergent issues, such as the H1N1 pandemic, in special populations.

ELIGIBILITY:
Inclusion Criteria:

* Health care encounter within prior year (for Veterans).
* Face to face contact with Veterans (for health care providers)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with spinal cord injury
  Comparison group of Veterans without SCI/D
  Health care providers in the SCI/D System of Care
  Infection control chiefs at VA facilities
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccination | One year/influenza season
Influenza non-vaccine infection control strategies | One year/influenza season
Veterans and health care providers attitudes and beliefs about H1N1 | One year/influenza season

CONTACTS AND LOCATIONS:
Overall Officials: Sherri L. LaVela, MPH MBA PhD, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States